CLINICAL TRIAL: NCT02048553
Title: Tablet-guided Versus Freehand (Tab-Guide) Ventriculostomy : Study Protocol to the Test Accuracy of Ventriculostomy in a Randomized Controlled Trial
Acronym: Tab-Guide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Sarrafzadeh Asita, Professor of Neurosurgery (Charité Berlin, Germany), University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05092013
Record Dates: First submitted 2013-09-04; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Hydrocephalus.
Keywords: ventriculostomy; complications in neurosurgery;catheter accuracy;
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet-guided (Experimental): Guide-assisted ventriculostomy.
  Interventions: Procedure: Freehand
- Freehand (Experimental): standard ventriculostomy.
  Interventions: Device: Tablet-guided ventriculostomy

INTERVENTIONS:
Device: Tablet-guided ventriculostomy — In patients of the treatment group, ventriculostomy will be performed using a mini-tablet-guided assistance based on preoperative CT imaging. Any patient meeting the inclusion criteria and not violating the exclusion criteria may participate in the TABGUIDE study and be randomized to either a guided or freehand ventriculostomy, thus defining the two distinct groups " guided " or " freehand ").
  Other Names: TABGUIDE
  Arms: Freehand
Procedure: Freehand — Patients in the control group will receive standard free-hand ventriculostomy using anatomical landmarks. The catheter may be placed for external drainage or internal (ventriculoperitoneal) shunting in both groups.
  Arms: Tablet-guided

SUMMARY:
Background: Despite the widespread use of external ventricular drainage, revision rates and associated complications are reported between 10-40%. Current available image-guided techniques using stereotaxis, endoscopy or ultrasound for catheter placements remain time-consuming techniques. Recently, a phone-assisted guide with high precision has been described. The development of an easy-to-use, portable, image-guided system could reduce the need for multiple passes and improve the rate of accurate catheter placement. This study aim to compare prospectively in a randomized controlled manner the accuracy of the freehand pass technique versus an an easy-to-use, portable mini-tablet-assisted guide for ventriculostomy catheter placement.

Methods/Design: This is a single center, prospective, randomized, trial with blinded endpoint (ventricle catheter tip location) assessment. Adult patients with the indication for ventriculostomy, as proven by computed tomography (CT), will be randomly assigned to the treatment group or the control group. In patients of the treatment group, ventriculostomy will be performed using a mini-tablet-guided assistance based on preoperative CT imaging. Patients in the control group will receive standard free-hand ventriculostomy using anatomical landmarks. The catheter may be placed for external drainage or internal (ventriculoperitoneal) shunting in both groups. The primary outcome measure is rate of correct placements of the ventricular catheter, defined as a score of 1 to 3 on grading system for catheter tip location on postoperative CT scan. Primary outcome will be determined by one of the authors (NS) blinded for treatment allocation. We aim to include 320 patients in 3 years.

Secondary Outcome Measures include 1) Frequency of placements required, 2) Frequency of completed placements within the ventricle of the perforated part of the tip of the catheter, 3) Frequency of very early and early shunt failures (revision of the ventricular drainage within 24 hours / within three weeks, 4) Frequency and Percentage of complications (procedure-related and nonsurgical) within three weeks, 5) Length of the trajectories from the dura level to the foramen of Monroe, the angle in the coronal plane towards midline (a) and towards the target (b) at the respective entry point, 6) ventricle size (the frontal occipital horn ratio (FOHR) and the width of the lateral ventricle in the coronal plane between the medial wall of the corpus callosum and the septum), 7) Differences (angles, distance of catheter tip from target) on the tablet-guided planned and postoperative trajectory on control computer tomography within 48 hrs (CT).

Discussion: Here, we present the study design of a single center prospective randomized controlled trial to investigate whether tablet-guided application ventriculostomy is superior to the standard free hand technique. The strengths of this study are: 1. the prospective, randomized interventional character testing a new easy-to handle guided versus free-hand ventricular catheter placement, and 2. the power calculation is based on catheter accuracy using an available grading system for catheter tip location and calculated with use of recent study results of our own population, supported by data from prominent studies.

DETAILED DESCRIPTION:
Methods Design The Tablet-guided versus freehand ventriculostomy (TABGUIDE) study will be performed as a 2-arm randomized controlled single-center trial to compare an intervention group using a guided placement of a ventricular catheter to a control group receiving standard (free-hand) ventriculostomy with blinded endpoint (catheter tip location) assessment.

Setting The present study is in compliance with the Helsinki Declaration. The protocol of this study was approved by the Ethics Committee on Human Research (CER) of the Medical Faculty of the University of Geneva, Switzerland (reference number: CER 13-175). At the planned start of the study at 01. March 2014, the study center will start randomization.

Randomization The randomization will start as soon as possible after consent to the study has been obtained. Any patient meeting the inclusion criteria and not violating the exclusion criteria may participate in the TABGUIDE study and be randomized to either a guided or freehand ventriculostomy, thus defining the two distinct groups " guided " or " freehand ". Online randomization will be performed by the treating physician in the study center using permuted blocks, to ensure an equal number of patients in both study arms.

Interventions - Surgical technique

The study is conducted in the neurosurgical department of a swiss single center university hospital in adult patients with indication for a ventricular drainage (such as hydrocephalus, slit ventricles, pseudotumor cerebri). Data management and monitoring will be performed by the Geneva study center and statistical analysis by one of the authors (NS).

For guidance, an easy-to handle instrument assisted by a mini-I-pad (mini-tablet)application software (Apple Inc.) is used in order to achieve precise placement of ventricular catheters on an every-case basis. The catheter may be placed for external drainage or internal (ventriculoperitoneal, VP) shunting.

For patients in the guided group, catheter placement is performed in the operating theatre during anesthesia under routine sterile conditions and antibiotic prophylaxis. The phone-assisted technique used for guided placing of a ventricular catheter through an burr hole has been previously described in detail. The only difference is the use of a easy-to-use portable mini-tablet available for all neurosurgeons instead of a phone. In brief, the patient is positioned and draped in typical sterile fashion for ventriculostomy (if necessary enlarged for shunt placement). Using a standard adult perforator (14 mm; AESCULAP, Germany), a frontal burr hole is made.

The guiding instrument consists of a base with three pins in order to be rigidly placed on the bone surface over the burr hole. A semicircular guide rod is mounted to the base in which an angle scale is engraved. Within the guide rod, a tube can be individually adjusted in one orientation at different angulations with a range from -600 to 600. Different tubes are designed with inner diameters of 2, 2.5, and 3 mm in order to guide catheters at different sizes. At the respective angle adjustment, the tube is fixed to the guide rod by a mounting screw. The base is opened at one side to enable the view or insert any instrument towards the lower opening of the tube. The guiding tool is positioned parallel to the midline along the engraved linear markings on the base of the instrument. Thereby, a rectangular insertion towards the sagittal convexity and an individual insertion angle towards the coronal tangent at the entry point can be established via the tube.

After dura opening, once the appropriate trajectory is chosen, the catheter is inserted according to the precalculated insertion angle. After tactile feedback of entering the ventricle, the stylet is removed. Cerebrospinal fluid (CSF) drainage ensures that the ventricular catheter is sufficiently in place. Catheters deemed to be suboptimally placed are repositioned when necessary. We rely on length markings on the ventricular catheter and, when possible, flow through the distal catheter to ensure the catheter has not been moved after fixation on the skin and is continuing to provide a conduit for CSF. The remainder of the possibly following shunt procedure or connection to a Ommaya reservoir was performed with standard techniques.

The classical freehand technique uses anatomical landmarks and the catheter is placed in the anterior horn of the lateral ventricle through a burr hole just anterior to the coronal suture in the pupillary line (at the level of Kocher's point, a point on the surface of the cranium 2.5 cm from the midline and 1 cm anterior to the coronal suture). The target is the ipsilateral frontal horn just anterior to the foramen of Monroe to avoid the chorioid plexus. The right nondominant side is preferred. The catheter is directed freehand using external landmarks in the coronar plane towards the ipsilateral medial canthus and in the sagittal plane through the external auditory meatus. A post-procedural CT scan of the brain is performed within 24 hours as part of standard care for postoperative control or earlier in case of postoperative CSF drainage problems.

Mini-Tablet application Regular digital imaging (DICOM) viewing software, commonly used in clinics, to evaluate radiological imaging, integrates simple measurement tools (e.g. distance or angle measurements). This technique is used to define a trajectory with an entry point at the frontal paramedian convexity towards the foramen of Monroe in a coronal section. Then, measurements can be taken to determine the angle between the trajectory and the respective tangent at the entry point on the skull surface. An I-Phone (Apple Inc., USA) software application available is used, importing anonymous imaging material. This image should be a coronal section with the lateral ventricles shown at the level of the anterior commissure. The next step is to define a paramedian entry point on the surface of the skull by tapping the finger on the respective spot. Then, the two feet are virtually placed on the skull surface. A rectangular trajectory orientation of the tube is then shown as a dotted line and can be shifted if necessary. The angle deviation from a rectangular insertion is then given by the software as a value. In addition, the finger may be placed on the target within the ventricle, and the length of the catheter will be given as distance value. As alternative, the CT scan (at the level : coronal section with the lateral ventricles shown at the level of the anterior commissure) can be photographed and used for angle calculations.

Consent procedure Patients capable of consenting will be informed about the study details themselves and may or may not agree to participate. If the patient or his/her legal representative refuses consent after inclusion by advice of an independent physician, the patient's further study participation is no longer possible. In this case, however, the patient or his/her legal representative is asked to give consent for evaluation of already acquired data. The detailed explanation of the study to the patient, legal representative has to be carried out using appropriate explanations and words depending on the previous medical knowledge of the respective person and her/his level of education. During the explanations, the respective person will be asked on a regular basis if she/he understands the conveyed information and if any questions have arisen. In addition to these verbal explanations the patient/legal representative will be given a leaflet containing the study details. After reading the leaflet the respective person will be given as much time as she/he demands for the decision on study participation.

This study evaluates the outcome of an intervention performed often in an emergency situation. Since approximately half of patients will not be able to give informed consent at admission, the informed consent procedure for this study will be delayed in a so-called emergency procedure. If neither the patient is capable of giving informed consent nor a family representative (informed consent) is available in due time, an independent neurosurgeon not involved in the patient's treatment nor in the trial may be asked for study approval. This option was introduced into the consent procedure because data on smart-phone guided ventriculostomy suggest a potentially beneficial effect of the measure for the patient - however performed in a small group of 35 patients. Therefore it shall not be categorically withheld from patients who are not capable of deciding whether to participate in the study or not and who do not have a legal representative. As soon as a legal representative / family representative is available and/or the patient is capable again to consent to the study, he or she must be asked to give informed consent.

Sample Size Analysis Sample size analysis estimates (hit and miss rates) were based on the results of observational studies. In a recent single center study of our group on the accuracy of ventricular catheter placement, using anatomic landmarks versus neuronavigation or CT-laser guidance, ventricles were hit in 69.2% of catheter insertions (31% miss rate) using anatomical landmarks (non-assisted), as compared to 82.3% with the use of guidance (neuronavigation or CT-guidance, p=0.043) (submitted data). The placements that were non-assisted were significantly more likely to be placed extraventricularly than those using guidance (OR 3.73, 95%, Confidence Interval (CI) 1.24, 11.19, p=0.019). Given data from other retrospective studies on ventricular catheters (in the context of ventricular-peritoneal shunts), similar rates between 25-45%4-7 of malpositioning are described.

To detect a decrease in the incidence of malpositioning from 35% to 20, 151 patients in each of the two study arms are needed to gain a power of 80%, using an alpha error of 5%. The final planned study size is to include and randomize 302 patients.

Data Management Data specified in the trial protocol will be documented in the patient's digital records. Additional clinical data are available from the electronic patient files. The investigating physician is responsible for appropriate completion of the form. The authors (AS, NS) are responsible for data base development, data acquisition, data storage, and validation. Data validation includes controls of completeness, consistence and plausibility of the data documented in electronic dossier using a query system between data management and investigating physician.

Adverse events (AE) and severe adverse events (SAE) The term " adverse event " (AE) describes any sign, symptom, syndrome or any disease 1. Occurring newly in a trial participant after consent to the trial and 2. Being of particular interest for the assessment of the disease or the security of the therapeutic concept. Any AE is documented in the electronic file of the patient.

Definition of Adverse Events (AE):

1. - Impairment of the general condition of the patient,
2. - Physical injury, including falls,
3. - Infection other than wound infection, sepsis or SIRS,
4. - Intracranial bleeding in the proximity of the ventricular catheter,
5. - Wound infection or dehiscence at the emersion site of the ventricular catheter,

7 - Newly occurred neurological deficit, 8 - Arterial or venous thrombosis, 9 - Any suspicious findings that may have relationship to the study.

Definition of Serious Adverse Events (SAE):

10 - Fatal events / Death, 11 - Any Life-threatening condition, 12 - Disabling or incapacitating events, 13- Events that require prolongation of hospitalization, 14 - Required intervention to prevent permanent impairment.

Relation (as cause or result) to other AE/SAE:

0 - No, 1 - Possible (give brief description), 2 - Yes (give brief description).

Investigator's estimation of the severity of the problem to the study or study device (fill in only, if AE/SAE is or might be related to study) 1 - Mild, 2 - Severe, 3 - Life Threatening.

Investigator's recommendation to change the protocol, informed consent or assent form 0 - No, 1 - Yes (give brief description).

Outcome of AE or SAE (until discharge)

1 - Full recovery, 2 - Permanent deficit, 3 - Not yet fully recovered, 4 - Not known.

Reporting & Statistical Analysis The reporting of this trial will conform to the reporting guidelines outlined in the CONSORT statement of 2010. The statistical analysis will be by intention-to-treat. The occurrence of the primary outcome, number and frequency of correct ventriculostomy, will be compared between the two randomization groups. The secondary outcome analyses will compare the above described variables between randomization groups. Subgroup analyses will be performed to evaluate whether other parameters such as age, ventricle size, diagnosis or experience of the surgeon may influence the results. Data are presented as mean and standard deviation or as median with 25/75 percentiles. Stata version 11.2 (College Station, Texas) will be used for all analyses.

Interim analyses This trial will follow a group sequential design, with 2 stop-points (interim and final analysis). The trial will stop if efficacy rules are met. The endpoints assessed at the first stop-point will be based on primary outcomes and adverse events. The first will be the interim analysis will occur after the accrual of 50 patients in each arm (100 total) thus representing approximately 1/3 of trial accrual. For the efficacy stop-point, a p-value of 0.001 at interim and 0.05 at final analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older,
* Indication for a ventricular drainage (such as hydrocephalus, slit ventricles, pseudotumor cerebri).

Exclusion Criteria:

* Pregnancy,
* Concurrent participation in another interventional trial (participation in an observational trial is not an exclusion criteria),
* postoperative imaging not to be performed,
* frontal burr hole not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and Percentage of correct placements of the ventricular catheter. | Assessed on postoperative cranial computer tomography, performed within 48 hours post intervention.
  Table 1. Grading system for catheter tip location Grade / Accuracy of placement / Location of catheter tip
  1. Optimal/adequate Ipsilateral frontal horn, including tip of third ventricle
  2. Suboptimal in noneloquent tissue Controlateral frontal horn or lateral ventricle/corpus callosum/interhemispheric fissure
  3. Suboptimal in eloquent tissue Brainstem/cerebellum/internal capsule/basal ganglia/thalamus/occipital cortex/basal cisterns
Frequency and Percentage of acute ventricular revisions. | 7 days
  2) Frequency and Percentage of acute ventricular revisions (within 1 week for an improperly-placed catheter). Assessment is performed by a blinded investigator of the study.

SECONDARY OUTCOMES:
Frequency of placements required. | During intervention.
  1) Frequency of placements required.
Frequency of correct placement. | on postoperative cranial computer tomography with 48 hrs post intervention.
  2) Frequency of completed placements within the ventricle of the perforated part of the catheter,
Frequency of very early and early shunt failures | within 24 hours / within the hospital stay
  3) Frequency of very early and early shunt failures (revision of the ventricular drainage within 24 hours / within three weeks,
Frequency and Percentage of complications | From intervention to discharge.
  4) Frequency and Percentage of complications (procedure-related and nonsurgical) within three weeks,
Length of the trajectories from the dura level to the foramen of Monroe | Evaluated on postoperative cranial computer tomography with 48 hrs post intervention.
  5)Length of the trajectories from the dura level to the foramen of Monroe, the angle in the coronal plane towards midline (a) and towards the target (b) at the respective entry point,
ventricle size | Evaluated on postoperative cranial computer tomography with 48 hrs post intervention.
  ventricle size (the frontal occipital horn ratio (FOHR) and the width of the lateral ventricle in the coronal plane between the medial wall of the corpus callosum and the septum),
Differences on the planned and postoperative trajectories. | Evaluated on postoperative cranial computer tomography with 48 hrs post intervention.
  Differences (angles, distance of catheter tip from target) on the tablet-guided planned and postoperative trajectories.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neurosurgery, Geneva University Hospitals, Geneva Neuroscience Center, Faculty of Medicine, University of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Sarrafzadeh A, Smoll N, Schaller K. Guided (VENTRI-GUIDE) versus freehand ventriculostomy: study protocol for a randomized controlled trial. Trials. 2014 Dec 5;15:478. doi: 10.1186/1745-6215-15-478. PMID 25480528